CLINICAL TRIAL: NCT05775523
Title: A Prospective, Non-interventional (NIS), Long-term, Post-Authorisation Safety Study (PASS) of Patients Treated With Lonapegsomatropin
Brief Title: A Post-Authorisation Safety Study (PASS) of Patients Treated With Lonapegsomatropin
Acronym: SkyPASS
Status: Recruiting | Type: Observational
Sponsor: Ascendis Pharma Endocrinology Division A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Other Study IDs: ASND0033
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Growth Hormone Deficiency
Keywords: Human Growth Hormone; hGH; rhGH; GHD; Long Acting Growth Hormone; Lonapegsomatropin; Prodrug; Growth Failure; Growth Hormone Replacement Therapy; Sustained Release Growth Hormone; Growth Hormone Deficiency; TransCon hGH; Skytrofa; SkyPASS
MeSH Terms: conditions — Dwarfism, Pituitary; Failure to Thrive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients on SKYTROFA (Lonapegsomatropin)Treatment: SKYTROFA (Lonapegsomatropin) administered once-weekly by subcutaneous injection
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — No intervention

SUMMARY:
The goal of this study is to further characterise the potential long-term safety risks of lonapegsomatropin in patients treated with lonapegsomatropin under real-world conditions in the post-marketing setting.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients with GHD who are on treatment with lonapegsomatropin
* Patients being clinically managed in Europe or the USA
* Appropriate written informed consent/assent as applicable for the age of the patient
* Patients willing to comply with follow-up requirements of the study

Exclusion Criteria:

* Patients participating in any interventional clinical trial for short stature
* Patients being treated with a GH or IGF-1 therapy, other than lonapegsomatropin, at enrollment
* Patients for whom treatment with lonapegsomatropin is contraindicated
* Patients with closed epiphyses
* Patients with active malignant tumours
* Patients under antitumour therapy within the past 12 months prior to instituting GH therapy
* Hypersensitivity to somatropin or any of the excipients in lonapegsomatropin

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from centres in Europe and the USA will be eligible for enrollment into the study.
  Patients may be enrolled in the study if they are on treatment with lonapegsomatropin. The decision to treat the patient with lonapegsomatropin will be made prior to and independently of the decision to invite the patient to enroll into the study. Both patients naïve to GH treatment and patients previously treated with GH therapy will be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2033-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of neoplasms (benign, malignant and unspecified) | 5 years
Occurrence of type 2 diabetes mellitus | 5 years

SECONDARY OUTCOMES:
Occurrence of renal, hepatic, immunologic and neurologic adverse events | 5 years
Occurrence of medication errors in patients treated with lonapegsomatropin | 5 years
  Frequency and type of medication errors as reported by treating physician
Insulin-like Growth Factor-1 (IGF-1) response to lonapegsomatropin therapy | 5 years
  IGF-1 level (ng/mL)
Insulin-like Growth Factor-1 (IGF-1) response to lonapegsomatropin therapy | 5 years
  IGF-1 Standard Deviation Score (SDS)
Compare the occurrence of neoplasms (benign, malignant and unspecified) in patients treated with lonapegsomatropin with historical data from literature | 5 years
Compare the occurrence of type 2 diabetes mellitus in patients treated with lonapegsomatropin with historical data from literature | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Ascendis Pharma A/S
Locations (26):
- United States (26):
  - Ascendis Investigational Site, Phoenix, Arizona
  - Ascendis Investigational Site, Orange, California
  - Ascendis Investigational Site, Sacramento, California
  - Ascendis Investigational Site, San Francisco, California
  - Ascendis Pharma Investigational Site, Centennial, Colorado
  - Ascendis Investigational Site, Washington D.C., District of Columbia
  - Ascendis Investigational Site, Orlando, Florida
  - Ascendis Investigational Site, Tampa, Florida
  - Ascendis Investigational Site, Sandy Springs, Georgia
  - Ascendis Investigational Site, Boise, Idaho
  - Ascendis Investigational Site, Indianapolis, Indiana
  - Ascendis Investigational Site, Iowa City, Iowa
  - Ascendis Investigational Site, Louisville, Kentucky
  - Ascendis Investigational Site, Minneapolis, Minnesota
  - Ascendis Investigational Site, Las Vegas, Nevada
  - Ascendis Investigational Site, Lebanon, New Hampshire
  - Ascendis Investigational Site, Manchester, New Hampshire
  - Ascendis Investigational Site, Morristown, New Jersey
  - Ascendis Investigational Site, New Hyde Park, New York
  - Ascendis Investigational Site, Cincinnati, Ohio
  - Ascendis Investigational Site, Portland, Oregon
  - Ascendis Investigational Site, Columbia, South Carolina
  - Ascendis Investigational Site, Dallas, Texas
  - Ascendis Investigational Site, El Paso, Texas
  - Ascendis Investigational Site, Norfolk, Virginia
  - Ascendis Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No